CLINICAL TRIAL: NCT01329120
Title: Short and Long-term Effects of Surgical Repair of Pectus Excavatum and Pectus Carinatum - A Questionnaire Study of Persistent Post-surgical Pain, Health-related Quality of Life, Patient Satisfaction, and Aesthetic Outcome
Brief Title: Short and Long-term Effects of Surgical Repair of Pectus Deformities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MIRPEX-1
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2012-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pectus excavatum: Patients who has undergone minimally invasive repair of pectus excavatum
  Interventions: Procedure: Minimally invasive repair of pectus excavatum
- Pectus carinatum: Patients who has undergone open surgical repair of pectus carinatum
  Interventions: Procedure: Open surgical repair of pectus carinatum

INTERVENTIONS:
Procedure: Minimally invasive repair of pectus excavatum — Minimally invasive surgical technique basically consisting of inserting one or more convex steel bars under the sternum through small bilateral incisions in the thoracic wall
  Other Names: Nuss procedure
  Groups: Pectus excavatum
Procedure: Open surgical repair of pectus carinatum — Open surgical removal the affected cartilages bilaterally and the excess cartilage over the sternum
  Other Names: Ravitch procedure
  Groups: Pectus carinatum

SUMMARY:
A large number of institutions have reported their early results with minimally invasive repair of pectus excavatum and open repair of pectus carinatum, but only few have addressed the outcomes relevant to the concerns of the patients and even fewer have reported long-term results following bar removal. Even fewer studies have investigated the prevalence and characteristics of long term persistent post-surgical pain following surgical repair of pectus deformities. The reasons as to why acute postoperative pain in some patients persists and becomes chronic whereas in others the pain dies down shortly after wound healing are largely unknown, and why some patients complain of loss of sensibility in wide regions of their chest following surgery also remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Minimally invasive repair of pectus excavatum from 2001 throughout 2010.
* Open surgical repair of pectus carinatum from 2001 throughout 2010.

Exclusion Criteria:

* Not being able to fill in detailed questionnaires in Danish

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients referred to the Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby for the purpose of pectus deformity repair from January 1, 2001 to December 31, 2010 are invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Persistent post-surgical pain | At least 4 months following surgery
  Persistent post-surgical pain is in this study defined as pain developing after pectus surgery and lasting for at least 4 months. Other causes of pain (e.g. infection and malignancy) and pain continuing from a pre-existing pain problem will be excluded.
  Persistent post-surgical pain present at time of the study will be assessed by means of a specifically developed questionnaire including items from the Danish translation of the Brief Pain inventory (BPI-short form) and the Danish translation of the short version of the McGill Pain Questionnaire (SF-MPQ).

SECONDARY OUTCOMES:
Health related quality of life | At least 4 months following surgery
  Health-related quality of life (HRQol) will be assessed by means of a validated Danish version of the Short-Form (36) Health Survey (SF-36)
Patient satisfaction | At least 4 months following surgery
  Satisfaction with the result of the deformity repair and the perceived impact of the correction on health-related quality of life is assessed by means of questions about the emotional and practical consequences of, and satisfaction with pectus repair.
Aesthetic outcome | At least 4 months following surgery
  In order to assess the surgical outcome following pectus repair in terms of aesthetic outcome more objectively, patients are encouraged to upload or e-mail a digital frontal image of their chests. Two thoracic surgeons, including the operating surgeon, and a research secretary are instructed to evaluate the breast symmetry, scars on the chest, and the overall cosmetic result of the repair.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Grosen, PhD Fellow, Principal Investigator — Aarhus University Hospital Skejby; Hans K Pilegaard, MD, Study Director — Aarhus University Hospital Skejby; Mogens Pfeiffer-Jensen, MD, PhD, Study Chair — Aarhus University Hospital, Aarhus Sygehus; Vibeke E Hjortdal, Prof., MD, PhD, Study Chair — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital, Skejby, Department of Cardiothoracic and Vascular Surgery, Aarhus, Denmark